CLINICAL TRIAL: NCT01661088
Title: A Phase II Study of Neoadjuvant FOLFIRINOX and FDR-Gemcitabine With Concurrent IMRT in Patients With Borderline Resectable Pancreatic Cancer
Brief Title: A Study of Neoadjuvant FOLFIRINOX and FDR-Gemcitabine With Concurrent IMRT in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.007; HUM 47389 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-07-24; First posted 2012-08-09 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: Neoadjuvant FOLFIRINOX; FDR-Gemcitabine; Concurrent; IMRT; Borderline Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Treatment (Experimental): Patients will receive FOLFIRINOX x 6 followed by IMRT concurrent with fixed dose rate (FDR)-gemcitabine (1g/m^2) on days 1, 8, 22, 29.
  Intensity-modulated radiotherapy (IMRT): The prescribed dose was 50.0Gy in 2.0Gy per fraction.
  Patients without metastatic disease will be offered surgical exploration.
  Interventions: Drug: FOLFIRINOX; Radiation: Intensity-modulated radiotherapy (IMRT); Procedure: Surgical Exploration

INTERVENTIONS:
Drug: FOLFIRINOX — Starting dose levels as following:
  Oxaliplatin 85mg/m2 intravenously over 120 minutes on day 1. Irinotecan 180mg/m2 intravenously over 90 minutes on day 1. NOTE: patients homozygous for the UGT1A1 (TA)7 promoter allele will be treated at an initial lower dose 140mg/m2 (please see Section 6.3.a) Leucovorin 400mg/m2 intravenously over 90 minutes on day 1. 5FU 400mg/m2 as bolus intravenous injection following leucovorin on day 1. 5FU 2,400mg/m2 infused intravenously as a continuous infusion over 46 hours following the bolus 5FU, beginning on day 1.
Radiation: Intensity-modulated radiotherapy (IMRT) — 50.0Gy in 2.0Gy per fraction
Procedure: Surgical Exploration — Patients without metastatic disease will be offered surgical exploration.

SUMMARY:
The investigators hypothesize that the combination of the FOLFIRINOX regimen (a combination of 5-fluorouracil, irinotecan and oxaliplatin chemotherapy) to provide maximal systemic disease control and FDR-gemcitabine chemotherapy with concurrent IMRT (Radiation therapy) to address local disease, will achieve a significant improvement R0 resection (Radiation oncology repeat surgeries) rate in borderline resectable (surgical) pancreatic cancer and enhance disease free and overall survival in this patient population.

DETAILED DESCRIPTION:
Gemcitabine has been the cornerstone of systemic therapy for pancreas cancer over this past decade. Recently, a combination of 5-fluorouracil, irinotecan and oxaliplatin (FOLFIRINOX) was reported to have significant efficacy in advanced pancreatic cancer. Preclinical data suggests synergy between irinotecan and 5FU as well as between oxaliplatin and 5FU. Results of a phase II trial in advanced disease were reported in 2005 demonstrating a 26% confirmed response rate and median overall survival of 10.2 months. A follow-up phase III trial comparing FOLFIRINOX with gemcitabine for patients <75 years of age with advanced pancreatic cancer was presented at ASCO 2010 revealing improvement in PFS (6.4 vs 3.3 months, p=<.0001) and improved disease control rate (CR+PR+SD) (70.2% vs 50.9%, p=.0003). The most notable result was an impressive improvement in median overall survival with FOLFIRINOX compared to gemcitabine (11.1vs 6.8 months, p-value = <.0001, HR=.57). The main toxicity was grade 3/4 neutropenia (45.7% vs 18.7%, p=.0001) and increased risk of febrile neutropenia (5.4% vs 0.6%, p=.009)31.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologic or histologic confirmation of carcinoma arising in the pancreas.
* Patients must be deemed to have borderline resectable disease with no radiologic evidence of distant metastatic disease prior to registration.
* Specifically, patients must have at least one designation of borderline resectable and no designation of unresectable disease.
* Patients must have a life expectancy of at least 12 weeks, a Zubrod performance status of < 1 and be willing and medically able to undergo surgical resection.
* Patients must have adequate organ function defined as follows: absolute neutrophil count of > 1500/mm3, platelets > 100,000/mm3, serum Cr < 1.5 mg/dl, total bilirubin < 2.0 mg/dl with relief of biliary obstruction if present (PTC tube or endobiliary stent).
* Patients must be free of other active systemic malignancy, ongoing infection, or any other serious uncontrolled, concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* Patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial due to the unacceptable teratogenic toxicity of abdominal radiation and cytotoxic chemotherapy.
* Patients must be aware of the investigational nature of the therapy and provide written informed consent.

Exclusion Criteria:

* Patients with neuroendocrine tumors are excluded.
* Active systemic malignancy, ongoing infection, or any other serious uncontrolled, concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* Patients with preexisting peripheral neuropathy > grade 2 are ineligible
* Pregnant or nursing women are ineligible.
* Patients must have no history of previous chemotherapy for pancreatic cancer or any abdominal radiation therapy.
* Patients may not have used any investigational agent within 4 weeks prior to enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2017-08-10 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Tran NH, Sahai V, Griffith KA, Nathan H, Kaza R, Cuneo KC, Shi J, Kim E, Sonnenday CJ, Cho CS, Lawrence TS, Zalupski MM. Phase 2 Trial of Neoadjuvant FOLFIRINOX and Intensity Modulated Radiation Therapy Concurrent With Fixed-Dose Rate-Gemcitabine in Patients With Borderline Resectable Pancreatic Cancer. Int J Radiat Oncol Biol Phys. 2020 Jan 1;106(1):124-133. doi: 10.1016/j.ijrobp.2019.08.057. Epub 2019 Sep 5. PMID 31494181

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: Patients received FOLFIRINOX x 6 followed by IMRT concurrent with fixed dose rate (FDR)-gemcitabine (1g/m^2) on days 1, 8, 22, 29.
  Intensity-modulated radiotherapy (IMRT): The prescribed dose was 50.0Gy in 2.0Gy per fraction.
  Patients without metastatic disease were offered surgical exploration.
Period: FOLFIRINOX
Arm/Group | Study Treatment
Started | 25
Completed | 21
Not Completed | 4
Period: IMRT With FDR Gemcitabine
Arm/Group | Study Treatment
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients That Underwent an R0 Resection
Description: To determine the frequency of achieving an R0 resection using a neoadjuvant regimen of FOLFIRINOX followed by IMRT concurrent with fixed dose rate (FDR)-gemcitabine in patients with borderline resectable pancreatic cancer. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Study Treatment
Number analyzed (Participants) | 25
percentage of patients | 52

2. Secondary Outcome: Median Progression-free Survival Time
Description: To estimate progression-free survival as a function of time from study enrollment. Progression is defined as at least a 20% increase in the LD (longest diameter) of the primary lesion or the appearance of one or more new lesions
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Treatment
Number analyzed (Participants) | 25
months | 13.1 [7.3 to 24.7]

3. Secondary Outcome: Median Overall Survival Time
Description: To estimate overall survival as a function of time from study enrollment.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Treatment
Number analyzed (Participants) | 25
months | 24.4 [12.6 to 40.0]

ADVERSE EVENTS:
Time Frame: 30 days post treatment
Arm/Group | Study Treatment
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment (N=25)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (14)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (15)
Platelet count decreased (Investigations) | 3 (5)
White blood cell decreased (Investigations) | 9 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT01661088/Prot_SAP_000.pdf